CLINICAL TRIAL: NCT02369887
Title: Bureau AIDS, TB, and STI, Thailand Ministry of Public Health
Brief Title: Evaluation of a Facility-based Test, Treat, and Prevent HIV Program Among Men Who Have Sex With Men and Transgender Women in Thailand
Acronym: PrEP
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Other Study IDs: Test and Treat PrEP
Record Dates: First submitted 2015-02-05; First posted 2015-02-24 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2021-10

CONDITIONS: PrEP Test and Treat
Keywords: MSM/TG who agree to start PrEP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective observational cohort study that aims to enroll a total of 2000 Thai MSM and TG at five health facilities in four provinces of Thailand. Each participant will be followed for 18 months. Baseline and historical rates of HIV testing/re-testing, initial CD4 counts, retention in care, and ART adherence at the study clinics, at the study clinics combined, and national data (if available) will be compared with rates after implementation of the Test and Treat strategy. Analysis will also include an assessment of HIV prevalence and incidence. This study will use similar objectives, indicators, and procedures as those used in an ongoing Test and Treat study by the Thai Red Cross AIDS Research Centre in three tertiary care hospitals, and a study to be conducted with PEPFAR Key Populations Implementation Science (KPIS) funding through United States Agency for International Development (USAID), in community-based centers, allowing comparison of uptake and follow-up of MSM and TG using the Test and Treat strategy in a variety of settings.

ELIGIBILITY:
Inclusion Criteria:

* Thai national
* Age >18 year
* Male or transgender women who reports anal intercourse with a man without using a condom at least one time in the past 6 months
* Not known to be HIV-infected
* Able to read and write Thai

Additional inclusion criteria for PrEP:

* A negative HIV test result
* No signs or symptoms of acute HIV infection (fever, sore throat, fatigue, rash, swollen glands, nausea, diarrhea, white spots in the mouth) during the previous month
* Creatinine clearance >60 ml/min
* No contraindication to PrEP medication

Exclusion Criteria:

• Participating in community-based Test and Treat study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thai nationals not known to be HIV-infected aged ≥18 years old who are men or transgender women who report unprotected anal sex with a man in the past 6 months and are eligible for the study.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Pre-Exposure Prophylaxis of HIV | 36 months
  Participants must be Thai MSM or TG, aged 18 years or older, who report unprotected anal sex with a man during the previous 6 months, can read and write Thai, and are not known to be HIV-infected. To receive PrEP, participants must have a negative HIV test result, no signs or symptoms of acute HIV infection during the previous month, a creatinine clearance result > 60 ml/min, and no contraindication to PrEP medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Disease Control (DDC), Ministry of Public Health (MOPH), Nonthaburi, Thailand

REFERENCES:
- [Derived] Suraratdecha C, Stuart RM, Manopaiboon C, Green D, Lertpiriyasuwat C, Wilson DP, Pavaputanon P, Visavakum P, Monkongdee P, Khawcharoenporn T, Tharee P, Kittinunvorakoon C, Martin M. Cost and cost-effectiveness analysis of pre-exposure prophylaxis among men who have sex with men in two hospitals in Thailand. J Int AIDS Soc. 2018 Jul;21 Suppl 5(Suppl Suppl 5):e25129. doi: 10.1002/jia2.25129. PMID 30033559